CLINICAL TRIAL: NCT06006195
Title: Investigating the Correlation Between Dysphagia Symptoms and Swallowing Muscle Groups by High-Resolution Pharyngeal Manometry With Impedance, Along With the Associated Nutritional Assessment
Brief Title: Investigating the Correlations Between Dysphagia Symptoms and Swallowing Muscle Groups by HRPM-I
Status: Not yet recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Principal Investigator, National Taiwan University Hospital
Other Study IDs: 202306130RINB
Record Dates: First submitted 2023-08-06; First posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Swallowing Contraction Strength

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with dysphagia symptoms
  Interventions: Other: patients with dysphagia symptoms
- patients without dysphagia symptoms
  Interventions: Other: patients without dysphagia symptoms

INTERVENTIONS:
Other: patients with dysphagia symptoms — patients with dysphagia symptoms examined by high resolution impedance manometry
  Groups: patients with dysphagia symptoms
Other: patients without dysphagia symptoms — patients without dysphagia symptoms examined by high resolution impedance manometry
  Groups: patients without dysphagia symptoms

SUMMARY:
Investigating the correlation between the dysphagia symptoms and swallowing muscle groups by high resolution pharyngeal manometry with impedance

DETAILED DESCRIPTION:
Backgrounds: Some patients would experience dysphagia symptoms before the elective surgery. These patients usually do not have a history of head and neck surgery or cerebrovascular diseases. They are common causes of dysphagia. The anesthetics and airway manipulation can exacerbate dysphagia. However, research is limited on the specific weak muscle groups in patients with dysphagia symptoms, as well as on the existence of associated malnutrition.

Aims: The Eating Assessment Tool (EAT-10) questionnaire will be used to assess dysphagia symptoms. A score of ≥4 on the EAT-10 indicates the presence of dysphagia symptoms, while a score of <4 indicates the absence. This study aims to (1) investigate which specific muscle groups are particularly weak in patients with dysphagia symptoms (EAT-10≥4); (2) to examine whether patients with dysphagia symptoms (EAT-10≥4) have poorer nutritional status than patients without dysphagia symptoms (EAT-10<4).

Methods: This is a cross-sectional study. The investigators will recruit patients undergoing elective orthopedic surgery on the lower extremities, with the age range of 18 to 90 years. On the day of admission, patients will be examined by the EAT-10 questionnaire for dysphagia symptoms. High-resolution pharyngeal manometry with impedance will be conducted to measure the functional of swallowing muscles. Additionally, patients will be given the Mini Nutritional Assessment (MNA) questionnaire (a total score of 30 points). The higher scores indicate the better nutritional status. The albumin level will also be collected. The bioelectrical impedance analysis will be used to measure the patients' body composition, specifically skeletal muscle mass.

ELIGIBILITY:
Inclusion Criteria:

* age from 20 to 80 years

Exclusion Criteria:

* bleeding tendency
* pregnancy
* heart failure
* chronic kidney disease

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients age from 20 to 80 years old without major organ dysfunction
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-08-28 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
UES peak pressure, mmHg | 10 to 15 minutes

IPD SHARING:
Plan to Share IPD: No
due to ethical problem